CLINICAL TRIAL: NCT00825851
Title: Effect of Smoking, Abstention and Nicotine Replacement Therapy on Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: The Danish Medical Research Council (Other)
Responsible Party: Copenhagen Wound Healing Center, Bispebjerg Hospital, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: smokaw_3
Record Dates: First submitted 2009-01-20; First posted 2009-01-21 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Wound Healing
MeSH Terms: interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- continuous smoking (Active Comparator): subjects smoke 20 cigarettes per day
  Interventions: Behavioral: Continuous smoking
- smoking cessation and NRT (Active Comparator): subjects quit smoking and use transdermal nicotine patch
  Interventions: Drug: Transdermal nicotine patch; Behavioral: Smoking cessation
- smoking cessation and placebo patch (Placebo Comparator): subjects quit smoking and use placebo patch
  Interventions: Drug: Placebo patch; Behavioral: Smoking cessation
- never smokers (No Intervention): subjects being never smokers and who refrain from smoking

INTERVENTIONS:
Drug: Transdermal nicotine patch — 15mg/16h + 10mg/16h to be used 24h
  Other Names: Nicorette patch
  Arms: smoking cessation and NRT
Drug: Placebo patch
  Arms: smoking cessation and placebo patch
Behavioral: Smoking cessation
  Arms: smoking cessation and NRT; smoking cessation and placebo patch
Behavioral: Continuous smoking — subjects smoke 20 cigarettes per day
  Arms: continuous smoking

SUMMARY:
The aim was to determine the wound healing capacity in healthy never smokers and smokers who continue to smoke, or quit smoking using transdermal nicotine patch versus placebo patch.

DETAILED DESCRIPTION:
Two wound healing models were applied: the excisional skin biopsy model to study wound histology and the suction blister model to study epidermal regeneration and skin transudate. In addition blood sampling was made to validate compliance to the study arms and to study systemic markers of collagen metabolism and oxidative stress. In addition, wound infections and wound ruptures were recorded post hoc as complications to the excisional skin biopsy model were not expected to occur.

ELIGIBILITY:
Inclusion Criteria:

* daily smokers smoking between 15-25 cigarettes per day and never smokers

Exclusion Criteria:

* chronic medical disease
* atopic dermatitis or other skin disease
* pregnancy
* menopause
* allergy to dressings or patches
* current or recent medication with corticosteroids or NSAID

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2000-08; Primary Completion 2000-12 (Actual); Study Completion 2001-01 (Actual)

PRIMARY OUTCOMES:
wound healing | 1, 4, 8, and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lars T Sorensen, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

REFERENCES:
- [Result] Sorensen LT, Karlsmark T, Gottrup F. Abstinence from smoking reduces incisional wound infection: a randomized controlled trial. Ann Surg. 2003 Jul;238(1):1-5. doi: 10.1097/01.SLA.0000074980.39700.31. PMID 12832959